CLINICAL TRIAL: NCT03315884
Title: Pilot Randomized Clinical Study of the Iliac Arteries and Common Femoral Artery With Stenting Supera and the Iliac Arteries With Stenting and Plasty of the Common Femoral Artery Effectiveness in Patients With the Iliac and CFA Segment Occlusive or Stenosis Disease (TASC C, D)
Brief Title: Pilot Randomized Clinical Study of the Iliac Arteries and Common Femoral Artery With Stenting and the Iliac Arteries With Stenting and Plasty of the Common Femoral Artery
Acronym: TASC CD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Meshalkin Research Institute of Pathology of Circulation (Network)
Collaborators: Abbott (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: NRICP112
Record Dates: First submitted 2017-10-17; First posted 2017-10-20 (Actual); Last update posted 2020-05-28 (Actual); Status verified 2020-05

CONDITIONS: Atherosclerosis of the Peripheral Arteries
Keywords: TASC C, D; CFA; Supera; iliac arteries; common femoral artery; plasty of the common femoral artery; stenting Supera
MeSH Terms: interventions — Stents; Transdermal Patch

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Iliac segment recanalization and stenting Iliac segment CFA (Experimental): Iliac segment recanalization and stenting Iliac segment Common Femoral Artery (CFA)
  Interventions: Procedure: Iliac segment recanalization, stenting and plastic Common Femoral Artery (CFA) patch
- Iliac segment recanalization, stenting and plastic CFA patch (Active Comparator): Iliac segment recanalization, stenting and plastic Common Femoral Artery (CFA) patch
  Interventions: Procedure: Iliac segment recanalization and stenting Iliac segment Common Femoral Artery (CFA)

INTERVENTIONS:
Procedure: Iliac segment recanalization and stenting Iliac segment Common Femoral Artery (CFA) — Retrograde femoral access. Brachial access. Standard endovascular access is performed under local anesthesia and affected arterial segment is visualized. Stenosis or artery occlusion is passed with hydrophilic guide. In case of occlusion transluminal or subintimal (often "mixed") artery recanalization is performed. To maximize the preservation of the affected artery initial patency, occlusion recanalization is performed by ante-and retrograde accesses. Then stenosis or occlusion predilation is performed with balloon catheter (balloon catheter diameter is smaller than the affected artery diameter for 1-2 mm). After control angiography stent is installed in the aorta-iliac area throughout the lesion (lesion diameter corresponds to the stenotic arteries diameter). In aorta-iliac zone balloon-expandable and self-expandable stents are used.
  Other Names: Endovascular intervention
  Arms: Iliac segment recanalization, stenting and plastic CFA patch
Procedure: Iliac segment recanalization, stenting and plastic Common Femoral Artery (CFA) patch — Standard access to the CFA is performed. Outflow ways and CFA capability for reconstruction are determined. The puncture of the general CFA (retrograde) is performed and the introducer 7Fr. is set. Recanalization of iliac artery occlusion. It is necessary to cross the iliac occlusion in a retrograde fashion first and secure aortic inflow before making the arteriotomy. An ipsilateral, a contralateral and a brachial approaches are used depending on the clinical situation. If the retrograde access to the aorta failed, you use the antegrade crossing of the iliac occlusion with no intention to reenter the lumen in the CFA. After the recanalization and balloon angioplasty of iliac artery we completed the procedure with endarterectomy of CFA, patch closure and iliac stenting. The preference is to perform endarterectomy and patch before iliac stenting because it can be difficult to access the true lumen in a difficult CFA lesion. Controlling angiography were performed. Closing approach.
  Other Names: Hybrid Intervention
  Arms: Iliac segment recanalization and stenting Iliac segment CFA

SUMMARY:
According to the recommendations of the Inter-Society Consensus for the Management of Peripheral Arterial Disease (TASC II) statement and the Russian guidelines for limb ischemia treatment (2010), reconstructive surgery is preferred for type D lesions.

DETAILED DESCRIPTION:
According to the recommendations of the Inter-Society Consensus for the Management of Peripheral Arterial Disease (TASC II) statement and the Russian guidelines for limb ischemia treatment (2010), reconstructive surgery is preferred for type D lesions. Patients with type C lesions can be managed by either stenting or bypass surgery. Despite the fact that aorta-femoral reconstructions long-term results are better than the diffuse aorta-iliac lesions endovascular treatment results, the surgery risk is significantly higher than the endovascular surgery risk regarding criteria of mortality, complications, and return to normal activity.

All reports of iliac arteries stenosis percutaneous angioplasty indicate that the primary technical and clinical success rate exceeds 90%. The figure reaches 100% in the case of local lesions. The technical success of iliac arteries long occlusions recanalization reaches 80-85%. Improvement of endovascular equipment designed for the total occlusions treatment increases technical success of recanalization. The TASC II materials summarize the several large studies results which present the data on the operated segment artery patency at the level of 70-81% within 5-8 years of follow up. A large number of authors note the actuality of aortic-iliac type C and D segment lesions endovascular treatment recommendations revision according to the TASC II.

ELIGIBILITY:
Inclusion Criteria:

* Patients with occlusive lesions of C and D type iliac segment and CFA lesion, and with chronic lower limb ischemia (II-IV degree by Fontaine, 4-6 degree by Rutherford), age: 47-75 years old.
* Patients who consented to participate in this study.

Exclusion Criteria:

* Chronic heart failure of III-IV functional class by New York Heart Association (NYHA) classification.
* Decompensated chronic "pulmonary" heart
* Severe hepatic or renal failure (bilirubin> 35 mmol / l, glomerular filtration rate <60 mL / min);
* Polyvalent drug allergy
* Cancer in the terminal stage with a life expectancy less than 6 months;
* Acute ischemic
* Expressed aortic calcification tolerant to angioplasty
* Patient refusal to participate or continue to participate in the study

Ages: 47 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2017-12-01 (Actual); Primary Completion 2020-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Primary patency of the operated segment | during the whole period of observation. Observation is 24 month after surgery
  during the whole period of observation. confirmation of patency of the arterial ultrasound of the operated segment. Confirmation patency of artery 24 months after surgery using Multislice computed tomography angiography of the lower extremities

SECONDARY OUTCOMES:
Secondary patency of the operated artery restenosis | during the whole period of observation. Observation is 24 month after surgery
  during the whole period of observation. confirmation of patency of the arterial ultrasound of the operated segment. Confirmation patency of artery 24 months after surgery using Multislice computed tomography angiography of the lower extremities
reocclusion | during the whole period of observation. Observation is 24 month after surgery
  during the whole period of observation. confirmation of patency of the arterial ultrasound of the operated segment. Confirmation patency of artery 24 months after surgery using Multislice computed tomography angiography of the lower extremities
postoperative bleeding | in the early postoperative period. Surveillance is 30 days after surgery
  assessment of bleeding within 30 days after surgery. The identification of bleeding with physical examination and ultrasound.Considered bleeding requiring surgical intervention
hematoma | in the early postoperative period. Surveillance is 30 days after surgery
myocardial infarction | during the whole period of observation. Observation is 24 month after surgery
mortality | during the whole period of observation. Observation is 24 month after surgery
limb amputation | during the whole period of observation. Observation is 24 month after surgery
infection | during the whole period of observation. Observation is 24 month after surgery

CONTACTS AND LOCATIONS:
Locations (1):
- NRICP, Novosibirsk, Russia